CLINICAL TRIAL: NCT04536116
Title: EvaLuation De L'apport De L'Irm Virtuelle Sur La Qualité De La Prise En Charge Des Enfants En Irm
Brief Title: Virtual Reality As Anxiety Management Tool for Preparing Children for MR Exam
Acronym: LIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Servait Coralie, Radiology technician, Central Hospital, Nancy, France
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2019-A03072-55
Record Dates: First submitted 2020-08-05; First posted 2020-09-02 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2024-02

CONDITIONS: Claustrophobia
MeSH Terms: conditions — Claustrophobia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MRI simulation (Experimental): MRI simulation with a Virtual Reality headset
  Interventions: Device: Virtual Reality headset
- Standard medical care (No Intervention): Standard medical care

INTERVENTIONS:
Device: Virtual Reality headset — MRI simulation with a Virtual Reality headset
  Arms: MRI simulation

SUMMARY:
The access to MRI examination is limited due to the duration of the acquisitions, the noise and the narrow patient space of the device. A child can, therefore, be anxious, less cooperative and move more during the acquisition, affecting the quality of the examination and the medical diagnosis. General anesthesia or sedation, may be considered to obtain diagnostic quality examinations. Our hypothesis is that a scenario as close as possible to reality to prepare children before the MR exam could reduce their anxiety, improve the quality of the exams and reduce its duration.

The purpose of this study is to evaluate the effect of virtual reality on MRI exam preparation to reduce the anxiety of children (aged from 6 to 12 years) who are referred to their first MRI exam, as compared to the current practice.

ELIGIBILITY:
Inclusion Criteria:

* Child from 6 to 12 years old,
* Child who will have an MRI for the first time,
* Outpatient child,
* Child dependent on a parent affiliated to or beneficiary of a social security scheme,
* Child who has received age-appropriate information on the organization of the research,
* Child whose parents (or the only parent present with parental authority) have been fully informed about the organization of the research and have signed informed consent.

Exclusion Criteria:

* Conditions that not allow the realization of a virtual MRI sceanrio or not allow to respond the scales (epilepsy, mental disorders, language, ...),
* Child with a contraindication to performing an MRI,
* Child who has benefited from another MRI simulation system before ("IRM en Jeu" for instance)
* Child's opposition to participate.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2020-11-04 (Actual); Primary Completion 2023-10-18 (Actual); Study Completion 2023-10-18 (Actual)

PRIMARY OUTCOMES:
Anxiety | 2 hours
  Anxiety measurement before and after MRI by Visual Analogue Scale between 0 and 10

CONTACTS AND LOCATIONS:
Overall Officials: Coralie SERVAIT, PI, Principal Investigator — CHRU de Nancy
Locations (1):
- CHRU de Nancy, Vandœuvre-lès-Nancy, France